CLINICAL TRIAL: NCT05394909
Title: Treatment Of Giant Cell Arteritis Patients With Ultra-short Glucocorticosteroids And tociliZumab: Role of Imaging in a Observational Study
Brief Title: Ultra-short Glucocorticosteroids and Tocilizumab Therapy in GCA Patients
Acronym: TOPAZIO
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 186/2019/OSS
Record Dates: First submitted 2022-05-20; First posted 2022-05-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2022-05

CONDITIONS: GCA; TOCILIZUMAB; Glucocorticoids; PET
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tocilizumab 162Mg/0.9Ml Autoinjector — Patients will receive high-dose pulse intravenous methylprednisolone (500 mg ) for 3 consecutive days (Day 0-1-2) and subsequently will be treated weekly with Tocilizumab 162 mg s.c. for 52-weeks and then following according to SOC
  Other Names: methylprednisolone pulse 500 MG

SUMMARY:
The objective of our study is to evaluate the functional and morphological imaging variations at 24 and 52 weeks compared to baseline during TCZ-treatment and 6 months after the suspension of TCZ. We will also evaluate the variations of aortic dilatation during the study period using the PET/CT in comparison with an hystorical cohort of patients with LVV treated with GCs only and longitudinally followed at our rheumatology division.

DETAILED DESCRIPTION:
1. Trial Design Monocentric observational study, single arm, based on imaging of patients with active Large Vessel Giant Cell Arteritis (LV-GCA) , treated with Tocilizumab (TCZ) s.c. and with ultra-short glucocorticosteroids (GCs).
2. Duration of study per Subject 52 weeks of observation during standard of care (SOC) and 24 weeks of follow-up
3. Target Population Patients aged older than 50 years with active large vessel giant cell arteritis (LV-GCA) based on evidence of large vasculitis at imaging.

   Patients with active disease will be enrolled according to the following inclusion criteria:
   * PET/CT showing vascular FDG uptake ≥2 in at least one vascular district and at least one among
   * ESR >40 mm/h or CRP >10 mg/l
   * Cranial or systemic symptoms of GCA or symptoms of polymyalgia rheumatica (PMR)
4. Primary Objectives

   * To evaluate the functional and morphological imaging (PET and MRA scores) variations at 24, 52 and 76 weeks compared to baseline values.
   * To evaluate the proportion of patients with relapse free remission (RFR) at week 24, 52 and 76.
   * To assess agreement between of MRA and PET scores and physician-determined disease activity status.
5. Secondary Objectives

   * To evaluate if patients have a reduced risk of aortic dilatation compared with an hystorical cohort of patients with LVV treated with GCs only and longitudinally followed at our rheumatology division.
   * immunological effects of steroid and TCZ at baseline, after 3 days, at week 24, 52 and 76

ELIGIBILITY:
Inclusion Criteria

1. Patients aged older than 50 years with large vessel giant cell arteritis (LV-GCA)
2. PET/CT showing vascular FDG uptake ≥2 in at least one vascular district
3. ESR >40 mm/h or CRP >10 mg/l OR Cranial or systemic symptoms of GCA or symptoms of polymyalgia rheumatica (PMR)
4. Patient's written informed consent.

Exclusion Criteria

1. Use of more than 10 mg/day of prednisone (or equivalent) for more than 10 consecutive days in the previous three months
2. Rheumatic diseases (except for CPPD/chondrocalcinosis) other than GCA or polymyalgia rheumatica (i.e., RA, autoimmune connectivitides, other systemic vasculitides, a.o.)
3. Chronic use of systemic CS with inability, in the opinion of the investigator, to withdraw CS treatment at day 4 according to protocol
4. Evidence of significant and/or uncontrolled concomitant disease such as, but not limited to, cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine (in particular diabetes mellitus) or gastrointestinal disorders (including previous complicated diverticulitis) which, in the investigator's opinion, would preclude patient participation or impact the benefit-risk ratio
5. History of amaurosis fugax,visual loss or diplopia
6. Any condition or general state of health which, in the Investigator's opinion, would preclude participation in the study
7. Actual or recent myocardial infarction (within the last 3 months before screening visit)
8. Significant cardiac disease (NYHA Class III and IV), known severe chronic obstructive pulmonary disease (COPD) (FEV1 < 50% predicted or Functional dyspnea > Grade 3 on the MRC Dyspnea Scale) or other significant pulmonary disease
9. Uncontrolled disease (such as asthma, psoriasis or inflammatory bowel disease) where flares are commonly treated with oral or injectable corticosteroids
10. Known active infection of any kind, or any major episode of infection requiring hospitalization or treatment with i.v. anti-infectives within 4 weeks of baseline or completion of oral anti-infectives within 2 weeks before screening visit
11. History of deep space/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks before screening visit
12. Any surgical procedure, including bone/joint surgery within 8 weeks prior before screening visit or planned within the duration of the study
13. History of serious recurrent or chronic infection (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks before screening visit
14. Lack of peripheral venous access
15. Body weight > 150 kg or BMI > 35
16. Previous treatment with tocilizumab or any other biological agent within last 6 months before screening visit; Rituximab within 12 months before screening visit
17. Treatment with any investigational agent within 28 days of screening visit or 5 half-lives of the investigational drug (whichever is the longer)
18. History of severe allergic or anaphylactic reaction to any biologic agent or known hypersensitivity to any component of tocilizumab
19. Receipt of any vaccine within 28 days prior to screening visit (a patient's vaccination record and need for immunization prior to receiving tocilizumab/placebo must be carefully investigated)
20. Positive tests for hepatitis B surface antigen (HBsAg) or hepatitis C serology
21. Positive Quantiferon-TB® test for latent Tb without subsequent INH prophylaxis
22. Patients with active Tb which had to be treated for Tb within 2 years before the screening visit
23. Absolute neutrophil count (ANC) < 2.0 x 103/µL, white blood cells < 2.5 x 103/µL, platelet count < 100,000/ µL
24. Hemoglobin < 8.0 g/dL
25. Concentrations of serum IgG and/or IgM below 5.0 mg/mL and 0.40 mg/mL, respectively
26. Serum creatinine > 2.0 mg/dL (200 µmol/L)
27. Alanine aminotransferase (ALT) or aspartate amino-transferase (AST) > 1.5 times the upper limit of normal (ULN)
28. Total bilirubin > 1.5 times the upper limit of normal (ULN)
29. Triglycerides > 400 mmol/dL (non-fasted) or > 250 mmol/dL (fasted) at screening
30. Premenopausal status and nursing (definition of postmenopausal status: Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child-bearing potential)
31. Technical implants such as cardiac pacemakers (for MR-angiogram)
32. Claustrophobia (for MR-angiogram)
33. Known allergy against the contrast media (Multihance® or Dotarem® as alternative)
34. Evidence of malignant disease or malignancies diagnosed within the previous 5 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that have been excised and cured)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be focused on patients aged older than 50 years with active large vessel giant cell arteritis (LV-GCA) based on evidence of large vessel vasculitis (LVV) at imaging.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 24, 52 and 76 weeks variation of MRA grading of large vessel vasculitis | Baseline, 24, 52, 76 weeks
  To evaluate the morphological imaging (MRA scores) variations
Change from baseline at 24, 52 and 76 weeks variation of PET Vascular Activity Score (PETVAS) | Baseline, 24, 52, 76 weeks
  To evaluate the functional imaging (PET scores) variations
Change from baseline at 24, 52 and 76 weeks of the proportion of patients with relapse-free remission | Baseline, 24, 52, 76 weeks
  Remission will be defined as the absence of any clinical symptoms directly attributable to vasculitis with normalization of CRP/ESR and absence of new/worsened vascular damage at MRA and/or CT

SECONDARY OUTCOMES:
Variation of Aortic diameter at each time point | 24, 52, and 76 weeks
  Aortic dilatation will be defined by a diameter>40 mm in the ascending aorta, >40 mm in the thoracic descending aorta and >30 mm in the abdominal aorta. Any change of ≥5mm on serial CT will be considered significant aortic dilatation and significant progression of vascular damage.
Changes of concentrations of various cytokines in plasma and PBMC culture supernatants at each time point | Baseline, 3 days, 24, 52 and 76 weeks
  The levels of various cytokines in plasma samples and PBMC culture supernatants will be analyzed following activation with anti-CD3 / CD28 beads and lipolysaccharide (LPS).

CONTACTS AND LOCATIONS:
Overall Officials: carlo salvarani, MD, Principal Investigator — AUSL-IRCCS REGGIO EMILIA
Locations (1):
- Ausl-Irccs - S.C. Di Reumatologia, Reggio Emilia, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durmo R, Muratore F, Marvisi C, Cassone G, Ricordi C, Boiardi L, Mancuso P, Besutti G, Spaggiari L, Casali M, Croci S, Di Tommaso G, Leoni F, Fioroni F, Catanoso M, Giorgi Rossi P, Salvarani C, Versari A. Exploring total inflammatory vascular volume as a diagnostic and prognostic biomarker in giant cell arteritis. Rheumatology (Oxford). 2025 Nov 1;64(11):5863-5871. doi: 10.1093/rheumatology/keaf381. PMID 40650989
- [Derived] Muratore F, Marvisi C, Cassone G, Ricordi C, Boiardi L, Mancuso P, Besutti G, Spaggiari L, Casali M, Croci S, Durmo R, Versari A, Di Tommaso G, Catanoso M, Giorgi Rossi P, Salvarani C. Treatment of giant cell arteritis with ultra-short glucocorticoids and tocilizumab: results from the extension of the TOPAZIO study. Rheumatology (Oxford). 2025 May 1;64(5):3057-3062. doi: 10.1093/rheumatology/keae400. PMID 39150490
- [Derived] Muratore F, Marvisi C, Cassone G, Boiardi L, Mancuso P, Besutti G, Spaggiari L, Casali M, Croci S, Versari A, Giorgi Rossi P, Catanoso M, Costantini M, Galli E, Salvarani C. Treatment of giant cell arteritis with ultra-short glucocorticoids and tocilizumab: the role of imaging in a prospective observational study. Rheumatology (Oxford). 2024 Jan 4;63(1):64-71. doi: 10.1093/rheumatology/kead215. PMID 37195423